CLINICAL TRIAL: NCT05986565
Title: Pilot Trial of the FMF Connect Teacher Companion Website
Brief Title: Study of the Families Moving Forward Website Behavioral Intervention for Teachers of Students With Fetal Alcohol Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Christie Petrenko, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008481
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Fetal Alcohol Spectrum Disorders
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — Pyrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Website treatment (Experimental): This arm will receive access to the FMF teacher adapted website.
  Interventions: Behavioral: Families Moving Forward (FMF) Teacher adapted training
- delayed treatment control (Active Comparator): This arm will get the same intervention as the experimental arm delayed by 6 weeks.
  Interventions: Behavioral: Families Moving Forward (FMF) Teacher adapted training

INTERVENTIONS:
Behavioral: Families Moving Forward (FMF) Teacher adapted training — The FMF Connect Teacher Companion website is designed to offer teachers evidence-based education about FASD and strategies to support students with FASD. It is adapted from the FMF Program and FMF Connect, evidence based interventions to support caregivers of children with FASD. The FMF Program and FMF Connect aim to improve caregivers' efficacy and satisfaction as a parent, efficacy, attributions for their child's behavior, and the parent-child relationship.

SUMMARY:
The purpose of this study is to find out if the FMF Connect Teacher Companion website is acceptable and usable by teachers. The FMF Connect Teacher Companion website is a website for teachers adapted from the Families Moving Forward (FMF) Program. The FMF Program is an evidence-based intervention for caregivers of children with FASD. The study will determine if the a web page intervention is feasible and acceptable by looking at enrollment and retention of study subjects and acceptability of assessments.

ELIGIBILITY:
Inclusion Criteria:

* Be an educational professional currently actively employed in a school setting in the United States
* Be above the age of 18 years old
* Have direct, consistent contact with a student with a diagnosed fetal alcohol spectrum disorder (FASD) or confirmed prenatal alcohol exposure (PAE) between the ages of 5-12, (i.e. grades K to 5) in a special or general education classroom
* Have reliable access to the Internet
* Be able to consent for themselves

Exclusion Criteria:

* They are unable to read English
* They do not have direct, consistent contact with a student with a diagnosed FASD between ages 5-12 (e.g., substitute teacher, principal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kautz-Turnbull C, Carmichael Olson H, Coles C, Tapparello C, Love K, Luehmann A, Cole L, Toth S, Speybroeck E, Petrenko CLM. The Families Moving Forward Connect Teacher Companion website: Development and initial pilot randomized trial of an FASD-informed resource for teachers. Alcohol Clin Exp Res (Hoboken). 2025 Dec;49(12):2796-2809. doi: 10.1111/acer.70189. Epub 2025 Nov 12. PMID 41225288

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of a total of 145 people who completed the consent and screening process, 37 were deemed eligible and 108 were ineligible for the following reasons: 12 did not meet eligibility criteria, 21 were incomplete, and 75 were suspected fraudulent.
Period: Overall Study
Arm/Group | Website Treatment | Delayed Treatment Control
Started | 21 | 16
Baseline Surveys | 17 | 15
6-Weeks Surveys | 14 | 14
12-Weeks Surveys | 13 | 12
Completed | 13 | 12
Not Completed | 8 | 4
Not completed — Lost to Follow-up | 8 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Website Treatment | Delayed Treatment Control | Total
Number analyzed (Participants) | 21 | 16 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.57 (13.86) | 39.58 (8.82) | 41.85 (11.96)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 20 | 16 | 36
  Sex: Male | 0 | 0 | 0
  Sex: Unknown | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 16 | 35
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 15 | 33
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Knowledge About FASD From Baseline to 6 Weeks
Description: Teacher FASD knowledge will be measured using the "Fetal Alcohol Spectrum Disorder (FASD) Knowledge" survey. The survey scores range from 0-33 with higher scores indicating more knowledge about FASD.
Time Frame: baseline to 6 weeks
Population: Participants with data at 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Website Treatment | Delayed Treatment Control
Number analyzed (Participants) | 14 | 14
units on a scale
  Baseline | 15.50 (2.53) | 17.14 (2.45)
  6 weeks | 16.57 (3.54) | 17.14 (1.94)
Statistical Analysis 1: Comparison: Website Treatment vs Delayed Treatment Control; Test type: Superiority; p = 0.587, RMANOVA; 1

2. Primary Outcome: Change in Personal Efficacy Mean From Baseline to 6 Weeks
Description: Personal efficacy will be measured by the Personal Efficacy subscale of the Teaching Self-Efficacy Scale. This subscale has 5 items and ranges from 5-30, with higher scores indicating higher perceived personal efficacy.
Time Frame: baseline to 6 weeks
Population: participants with complete data on this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Website Treatment | Delayed Treatment Control
Number analyzed (Participants) | 11 | 12
units on a scale
  baseline | 23.36 (3.29) | 23.25 (2.53)
  6 weeks | 23.54 (3.24) | 23.08 (2.15)
Statistical Analysis 1: Comparison: Website Treatment vs Delayed Treatment Control; Test type: Superiority; p = 0.874, RMANOVA; 1

3. Primary Outcome: Change in Teaching Efficacy Means From Baseline to 6 Weeks
Description: Teaching efficacy will be measured by the Teaching Efficacy subscale of the Teaching Self-Efficacy Scale. This subscale has 5 items and ranges from 5-30, with higher scores indicating higher perceived teaching efficacy.
Time Frame: baseline to 6 weeks
Population: participants with complete data for this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Website Treatment | Delayed Treatment Control
Number analyzed (Participants) | 11 | 13
units on a scale
  baseline | 22.27 (3.13) | 22.67 (5.48)
  6 weeks | 21.83 (3.92) | 22.42 (5.38)
Statistical Analysis 1: Comparison: Website Treatment vs Delayed Treatment Control; Test type: Superiority; p = 0.946, RMANOVA; 1

4. Primary Outcome: Mean Difference in Sensory Seeking Attributions at 6 Weeks
Description: Sensory seeking attributions will be measured using the "Reasons for Children's Behavior" survey. This subscale has 5 items and scores range from 5-30, with higher scores representing higher endorsement of sensory seeking attributions.
Time Frame: 6 weeks
Population: participants with complete data on this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Website Treatment | Delayed Treatment Control
Number analyzed (Participants) | 13 | 13
units on a scale | 16.38 (5.84) | 14.00 (4.81)
Statistical Analysis 1: Comparison: Website Treatment vs Delayed Treatment Control; Test type: Superiority; p = 0.267, t-test, 2 sided; 24

5. Primary Outcome: Mean Difference in Sensory Avoiding Attributions at 6 Weeks
Description: Sensory avoiding attributions will be measured using the "Reasons for Children's Behavior" survey. This subscale has 5 items and scores range from 5-30, with higher scores representing higher endorsement of sensory avoiding attributions.
Time Frame: 6 weeks
Population: participants with complete data on this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Website Treatment | Delayed Treatment Control
Number analyzed (Participants) | 14 | 13
units on a scale | 19.36 (6.02) | 15.85 (7.39)
Statistical Analysis 1: Comparison: Website Treatment vs Delayed Treatment Control; Test type: Superiority; p = 0.187, t-test, 2 sided; df=25

6. Primary Outcome: Mean Difference in Task - Willful Attributions at 6 Weeks
Description: Task - willful attributions will be measured using the "Reasons for Children's Behavior" survey. This subscale has 3 items and scores range from 3-18, with higher scores representing higher endorsement of task - willful attributions.
Time Frame: 6 weeks
Population: participants with complete data on this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Website Treatment | Delayed Treatment Control
Number analyzed (Participants) | 14 | 12
units on a scale | 7.43 (2.87) | 7.08 (2.94)
Statistical Analysis 1: Comparison: Website Treatment vs Delayed Treatment Control; Test type: Superiority; p = 0.765, t-test, 2 sided; df=24

7. Primary Outcome: Mean Difference in Task - Ability Attributions at 6 Weeks
Description: Task - ability attributions will be measured using the "Reasons for Children's Behavior" survey. This subscale has 5 items and scores range from 5-30, with higher scores representing higher endorsement of task - ability attributions.
Time Frame: 6 weeks
Population: participants with complete data on this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Website Treatment | Delayed Treatment Control
Number analyzed (Participants) | 14 | 13
units on a scale | 20.71 (3.60) | 17.62 (4.54)
Statistical Analysis 1: Comparison: Website Treatment vs Delayed Treatment Control; Test type: Superiority; p = 0.060, t-test, 2 sided; df=25

8. Primary Outcome: Mean Difference in Disruptive Behavior Attributions at 6 Weeks
Description: Disruptive behavior attributions will be measured using the "Reasons for Children's Behavior" survey. This subscale has 5 items and scores range from 5-30, with higher scores representing higher endorsement of disruptive behavior attributions.
Time Frame: 6 weeks
Population: participants with complete data on this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Website Treatment | Delayed Treatment Control
Number analyzed (Participants) | 13 | 13
units on a scale | 12.08 (5.19) | 10.85 (6.77)
Statistical Analysis 1: Comparison: Website Treatment vs Delayed Treatment Control; Test type: Superiority; p = 0.608, t-test, 2 sided; df=24

9. Primary Outcome: Mean Difference in Emotional Support Attributions at 6 Weeks
Description: Emotional support seeking attributions will be measured using the "Reasons for Children's Behavior" survey. This subscale has 4 items and scores range from 4-24, with higher scores representing higher endorsement of emotional support seeking attributions.
Time Frame: 6 weeks
Population: participants with complete data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Website Treatment | Delayed Treatment Control
Number analyzed (Participants) | 14 | 13
units on a scale | 18.71 (3.75) | 17.92 (4.86)
Statistical Analysis 1: Comparison: Website Treatment vs Delayed Treatment Control; Test type: Superiority; p = 0.638, t-test, 2 sided; df=25

10. Primary Outcome: Mean Difference in Dysregulated Behavior Attributions at 6 Weeks
Description: Dysregulated behavior attributions will be measured using the "Reasons for Children's Behavior" survey. This subscale has 3 items and scores range from 3-18, with higher scores representing higher endorsement of dysregulated behavior attributions.
Time Frame: 6 weeks
Population: participants with complete data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Website Treatment | Delayed Treatment Control
Number analyzed (Participants) | 13 | 13
units on a scale | 10.31 (3.45) | 7.77 (3.61)

11. Primary Outcome: Mean Overall Quality of Website (Website Group Only)
Description: Overall quality will be measured using the Mobile Application Rating Scale - user version. Overall quality is a sum of the Engagement, Functionality, Aesthetics, and Information subscales. Each subscale represents a mean of items and ranges from 1 to 6. The overall total quality score is a sum of these scales and ranges from 4 to 24, with higher scores indicating higher overall quality.
Time Frame: 6 weeks
Population: participants with complete data for this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Website Treatment
Number analyzed (Participants) | 12
units on a scale | 16.88 (2.00)

12. Primary Outcome: Mean Subjective Quality of Website (Website Group Only)
Description: Subjective quality will be measured using the Subjective Quality subscale of the Mobile Application Rating Scale - user version. This subscale has 4 items in total. Each item is rated on a scale from 1 to 6 and the total score represents a mean across items, with higher scores indicating higher subjective quality.
Time Frame: 6 weeks
Population: participants with complete data on this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Website Treatment
Number analyzed (Participants) | 14
units on a scale | 3.70 (0.72)

13. Primary Outcome: Mean Perceived Impact of Website (Website Group Only)
Description: Perceived impact will be measured using the Perceived Impact subscale of the Mobile Application Rating Scale - user version. This subscale has 5 items in total. Items are rated on a scale from 1 to 6. Total scores represent a mean rating across items, with higher scores indicating higher perceived impact.
Time Frame: 6 weeks
Population: participants with complete data on this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Website Treatment
Number analyzed (Participants) | 14
units on a scale | 4.04 (0.77)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events teachers could include harm to self or others. However, these occurrences are unlikely to be a direct consequence of participation in the website intervention or study. These were not systematically assessed but procedures were in place to assess risk and respond appropriately if they arose.
Arm/Group | Website Treatment | Delayed Treatment Control
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/16
Other Adverse Events (participants affected / at risk) | 0/21 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT05986565/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT05986565/ICF_001.pdf